CLINICAL TRIAL: NCT00000271
Title: New Approaches to Cocaine Abuse Medications (A)
Brief Title: New Approaches to Cocaine Abuse Medications (A) - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3881; 5P50DA009236-18 (NIH)
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: Desipramine, cocaine, depression
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Depression | interventions — Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desipramine (Experimental): Participants were treated with desipramine, up to 300 mg per day. All patients received weekly individual manual-guided relapse prevention therapy.
  Interventions: Drug: Desipramine
- Placebo (Placebo Comparator): Participants were treated with matching placebo. All patients received weekly individual manual-guided relapse prevention therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desipramine — Participants were treated with desipramine, up to 300 mg per day, or matching placebo. All participants received weekly individual manual-guided relapse prevention therapy.
  Other Names: desmethylimipramine
  Arms: Desipramine
Drug: Placebo — Participants were treated with matching placebo. All participants received weekly individual manual-guided relapse prevention therapy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the effect of desipramine in cocaine abusers selected for major depression or dysthymia.

DETAILED DESCRIPTION:
This is a randomized, 12-week, double-blind, 'placebo-controlled trial of outpatients meeting DSM-III-R criteria for cocaine dependence and major depression or dysthymia (by SCID interview). Participants were treated with desipramine, up to 300 mg per day, or matching placebo. All patients received weekly individual manual-guided relapse prevention therapy. Weekly outcome measures included the Clinical Global Impression Scale, self-reported cocaine use and craving, urine toxicology, and the Hamilton Depression Scale.

ELIGIBILITY:
Inclusion:

1. Meets DSM-IV criteria for current cocaine dependence.
2. Used cocaine at least one day in the past month.
3. Currently meets DSM-IV criteria for Major Depression or Dysthymia.
4. Depressive disorder is either:

   1. primary (antedates earliest lifetime substance abuse or
   2. persistent during 6 months of abstinence in the past or
   3. at least 3 months duration in the current episode
5. Age 18-60.
6. Able to give informed consent and comply with study procedures.

Exclusion:

1. Meets DSM-IV criteria for past mania (i.e. bipolar disorder), schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse.
2. History of seizures.
3. History of allergic reaction to desipramine or imipramine.
4. Chronic organic mental disorder.
5. Significant current suicidal risk.
6. Pregnancy, lactation or failure in sexually active female patients to use adequate contraceptive methods.
7. Unstable physical disorders which might make participation hazardous such as hypertension, hepatitis or diabetes.
8. Coronary vascular disease as indicated by history or suspected by abnormal ECG or history or cardiac symptoms.
9. Cardiac conduction system disease as indicated by QRS duration >0.11.
10. Current use of other prescribed psychotropic medications within the last 2 weeks.
11. History of failure to respond to a previous adequate trial of desipramine or another tricyclic antidepressant.
12. Currently meets criteria for another substance dependence disorder (DSM-IV) other than nicotine, marijuana or alcohol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 1995-01 (Actual); Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Cocaine Use | Weekly over a 12 week period.
  Clinical Global Impression Scale, self-reported cocaine use and craving, urine toxicology.
Depression | Bi-weekly over a 12 week period.
  Hamilton Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Research Foundation for Mental Hygiene, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDowell D, Nunes EV, Seracini AM, Rothenberg J, Vosburg SK, Ma GJ, Petkova E. Desipramine treatment of cocaine-dependent patients with depression: a placebo-controlled trial. Drug Alcohol Depend. 2005 Nov 1;80(2):209-21. doi: 10.1016/j.drugalcdep.2005.03.026. PMID 15913920